CLINICAL TRIAL: NCT05793073
Title: Efficacy of an Antimicrobial Stewardship Intervention for Early Adaptation of Empirical Antibiotic Therapy in High-risk Neutropenic Patients
Brief Title: AMS Intervention for Early Adaptation of Empirical Antibiotic Therapy in High-risk Neutropenic Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Infectio01
Record Dates: First submitted 2023-03-16; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Neutropenia
Keywords: antibiotic; antimicrobial stewardship; hematological malignancy; febrile neutropenia
MeSH Terms: conditions — Neutropenia; Hematologic Neoplasms; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-intervention group
- Post-intervention group

SUMMARY:
Febrile neutropenia (FN) is a frequent and serious complication in patients with hematological malignancies undergoing intensive chemotherapy. The growth of antibiotic resistance is a major threat in high-risk neutropenic patients given that delay in introduction of appropriate empirical antibiotic therapy (EAT) in this population is associated with increased morbidity and mortality.

In 2013, the 4th European Conference on Infections in Leukaemia (ECIL-4) group published new guidelines, promoting early adaptation of EAT in stable afebrile patients, regardless of neutrophil count and expected duration of neutropenia. Despite these evidence-based guidelines, discontinuation and de-escalation strategies are not widely implemented in hematology departments. However, recent studies have found that early adaptation of EAT is safe and feasible and could lead to reduced antibiotic consumption.

In response to growing antibiotic resistance and low adherence to ECIL-4 guidelines in the hematology department in the center of Nice, the investigators have developed and implemented a multifaceted AMS intervention. This intervention aimed to improve the quality of febrile neutropenia management and to promote the adoption of early de-escalation and discontinuation strategies in high-risk neutropenic patients by our hematology team.

The aim of this before-after study was to assess the impact of a multifaceted AMS intervention, promoting early adaptation of empirical antibiotic therapy, on antibiotic consumption and clinical outcomes in high-risk neutropenic patients. Secondly, the investigators sought to assess the applicability and adherence to de-escalation and discontinuation strategies by the hematology team.

The primary endpoint was total antibiotic use during hospital stay, expressed as days of therapy (DOT). DOT was defined as the number of days that a patient received antibiotics regardless of the dose. Secondary endpoints included length of therapy (LOT), antibiotic-free days (AFD), 30-day mortality, ICU admission, Clostridium difficile infection and duration of stay. LOT was defined as the number of days that a patient received systemic antibiotic therapy, irrespective of the number of different antibiotics.

DETAILED DESCRIPTION:
INTRODUCTION

Febrile neutropenia (FN) is a frequent and serious complication in patients with hematological malignancies undergoing intensive chemotherapy. FN episodes are responsible for repeated and prolonged antibiotic therapy, leading to an increased risk of bacterial antibiotic resistance, Clostridium difficile infections, fungal infections and adverse drug events. The growth of antibiotic resistance is a major threat in high-risk neutropenic patients given that delay in introduction of appropriate empirical antibiotic therapy (EAT) in this population is associated with increased morbidity and mortality.

Excessive and inappropriate antibiotic use are major drivers of the growth of antibiotic resistance. Antimicrobial stewardship (AMS) interventions have therefore been introduced to optimize antibiotic use in order to decrease unintended consequences of antibiotic use, such as growing antibiotic resistance and excessive healthcare costs. AMS interventions often include various components, such as prescriber education, prospective audit and feedback as well as clinical decision support at the point-of-care.

In 2013, the 4th European Conference on Infections in Leukaemia (ECIL-4) group published new guidelines, promoting early adaptation of EAT in stable afebrile patients, regardless of neutrophil count and expected duration of neutropenia. Despite these evidence-based guidelines, discontinuation and de-escalation strategies are not widely implemented in hematology departments. However, recent studies have found that early adaptation of EAT is safe and feasible and could lead to reduced antibiotic consumption. However, some of these studies did not use a control group. Furthermore, some of these studies solely investigated the effets of one aspect of adaptation (i.e. de-escalation or discontinuation) or focused on specific clinical presentations or patient profiles. One interrupted time series study investigated the impact of de-escalation and discontinuation strategies on antibiotic consumption but found no significant difference in total antibiotic consumption.

In response to growing antibiotic resistance and low adherence to ECIL-4 guidelines in the hematology department in our center, the investigators have developed and implemented a multifaceted AMS intervention. This intervention aimed to improve the quality of febrile neutropenia management and to promote the adoption of early de-escalation and discontinuation strategies in high-risk neutropenic patients by our hematology team.

The aim of this before-after study was to assess the impact of a multifaceted AMS intervention, promoting early adaptation of empirical antibiotic therapy, on antibiotic consumption and clinical outcomes in high-risk neutropenic patients. Secondly, the investigators sought to assess the applicability and adherence to de-escalation and discontinuation strategies by the hematology team.

METHODS

Study population This study was conducted in the hematology department of a 1800-bed university teaching hospital in Nice, France during two 6-month periods. The hematology department is divided into two separate units: a 10-bed intensive care unit with laminar air flow rooms and a 16-bed conventional hospitalization unit.

During these periods, all patients admitted to the hematology department for intensive chemotherapy, with chemotherapy-induced neutropenia lasting 7 days or more, who experienced at least one febrile episode, were eligible for inclusion. Patients were excluded if they were younger than 18 years old or had chemotherapy-induced neutropenia for less than 7 days or received corticosteroids.

Design and implementation of AMS intervention The pre-intervention spanned from October 2019 to March 2020. During this period, if EAT was effective (i.e patient remained stable and apyrexia was obtained), no change to antibiotic regimen was made, discontinuation was not considered and de-escalation was rarely performed. During this period, the discontinuation of antibiotic therapy was solely determined by neutrophil recovery.

In early 2021, the investigators started to design a persuasive multifaceted AMS intervention, aimed to optimize the management of high-risk febrile neutropenia. The implementation of the intervention started on November 2nd 2021 and the implementation phase lasted one month. This intervention included the development of new local clinical guidelines in the form of visual decision algorithms, prompting early de-escalation and discontinuation of EAT, according to clinical and microbiological criteria. These decision algorithms were subsequently discussed with the hematology medical team and revised until they were agreed upon by both teams. These visual decision aids were then displayed in all medical offices of the hematology department. Educational meetings were held with residents and paramedical staff during the implementation period, providing an opportunity for all stakeholders to ask questions and to learn about the adaptation guidelines. Additionally, a patient-level review of all antibiotic prescriptions was conducted twice a week in the presence of the hematology medical team and the AMS team. Patient-specific recommendations regarding antibiotic therapy were provided by the AMS team based on clinical and microbiological data. Moreover, the AMS team offered day-to-day guidance via a specialist hotline.

The post-intervention phase started in December 2021 and lasted for the subsequent 6 months, until May 2022. During this period, clinical outcomes and adherence to clinical algorithms were prospectively assessed and face-to-face meetings were organized by the AMS team to provide feedback on progress of the intervention and to discuss opportunities for improvement with the hematology team.

Febrile neutropenia guidelines In November 2021, new clinical guidelines promoting early adaptation of EAT, based on local microbiological epidemiology, clinical and microbiological criteria and ECIL-4 guidelines, were introduced.

In line to guidelines, EAT with a beta-lactam agent was started as early as possible after onset of fever in neutropenic patients. During both periods, carbapenem use was restricted to patients with prior colonization or infection with ESBL-producing bacteria and in patients with septic shock. A single injection of aminoglycosides was administered in patients with sepsis or septic shock. An agent active against resistant Gram-positive (e.g. daptomycin, vancomycin or linezolid) was added in patients with suspected catheter-related infection, skin and soft tissue infection or severe mucitis, in patients with prior colonization or infection with methicillin-resistant Staphylococcus aureus (MRSA) as well as in patients with septic shock.

Without documented infection, EAT was discontinued after 72 hours in stable patients who had been afebrile for at least 48 hours, irrespective of neutrophil count or expected duration of neutropenia. In clinically or microbiologically documented infections, appropriate antibiotic therapy was continued for at least 7 days and until infection was microbiologically eradicated and clinical resolution was obtained and fever had resolved for at least 4 days.

If an anti-resistant Gram-positive agent was started based on focal clinical signs, its stopping was encouraged in stable patients who had been afebrile for at least 48 hours upon resolution of focal clinical signs. If EAT with carbapenem was started based on prior colonization or infection with resistant pathogens and no microbiological documentation was available, de-escalation was encouraged in stable patients who had been afebrile for at least 48 hours. If carbapenem or anti-resistant Gram-positives therapy was started in the context of septic shock and the patient had stabilized on treatment, without documented infection, no particular change was encouraged.

Data collection All individual data on the pre-intervention period was retrospectively collected by the AMS team by manual review of electronic health records (EHRs) while data on the post-intervention phase was prospectively collected. Data on patient demographics, comorbidities, hematological malignancies, colonization with multidrug-resistant (MDR) bacteria (i.e. MRSA or ESBL-producing bacteria), dates and reason for hospital stay, results of microbiological samples, were collected. All data on antibiotic use were also retrieved from EHRs and were then double checked for accuracy by the pharmacy department. Clinical outcomes, such as ICU admission and 30-day mortality, were also collected to assess for unintended consequences of early adaptation of EAT. The applicability of de-escalation and discontinuation strategies and clinician adherence to these strategies were also assessed by the AMS team individually for all FN episodes.

The primary endpoint was total antibiotic use during hospital stay, expressed as days of therapy (DOT). DOT was defined as the number of days that a patient received antibiotics regardless of the dose. When a patient received more than one antibiotic, more than one DOT was counted. Secondary endpoints included length of therapy (LOT), antibiotic-free days (AFD), 30-day mortality, ICU admission, Clostridium difficile infection and duration of stay. LOT was defined as the number of days that a patient received systemic antibiotic therapy, irrespective of the number of different antibiotics [24]. AFD were calculated by the difference between duration of neutropenia of stay and LOT. If duration of neutropenia was greater than LOT, AFD was measured as 0. The 30-day mortality was defined as death occurring within 30 days after the onset of neutropenia.

Statistical analysis Continuous variables are reported as median (interquartile range) and categorical variables as number (percentage). Continuous variables were compared using the Student's t-test, or when inappropriate the Mann-Whitney test. Categorical variables were compared using the Chi-2 test, or when inappropriate the Fisher's exact test. All tests were two-tailed and p values ≤ 0.05 were considered statistically significant. Univariate and multivariate logistic regression was performed to identify factors associated with clinician adherence to de-escalation and discontinuation strategies. Only variables with p values < 0.2 in the univariate analysis were included in the multivariate logistic regression model. Sample size was calculated using a power of 80% and an α value of 0.05. Based on preliminary results from our department, the mean DOT was assumed to be 29 days (standard deviation = 13.5 days) and a reduction of DOT by 25 % in the post-intervention period was considered significant. Based on these assumptions, a sample size of 55 per period was required. The open-source software R Foundation for Statistical Computing (Vienna, Austria) was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the hematology department for intensive chemotherapy, with chemotherapy-induced neutropenia lasting 7 days or more, who experienced at least one febrile episode, were eligible for inclusion.

Exclusion Criteria:

* Younger than 18 years old
* Had chemotherapy-induced neutropenia for less than 7 days or received corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with febril neutropenia due to intensive chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Total antibiotic use during hospital stay, expressed as days of therapy (DOT) | 31 months
  DOT was defined as the number of days that a patient received antibiotics regardless of the dose. When a patient received more than one antibiotic, more than one DOT was counted.

SECONDARY OUTCOMES:
Total antibiotic use during hospital stay, expressed as days of therapy (LOT) | 31 months
  LOT was defined as the number of days that a patient received systemic antibiotic therapy, irrespective of the number of different antibiotics
Antibiotic-free days (AFD) | 31 months
  AFD were calculated by the difference between duration of neutropenia of stay and LOT. If duration of neutropenia was greater than LOT, AFD was measured as 0.
30-day mortality rate | 31 months
  The 30-day mortality was defined as death occurring within 30 days after the onset of neutropenia. Number of deaths among all hospital stays included during the study period.
ICU admission rate | 31 months
  Number of ICU admission among all hospital stays included during the study period.
Clostridium difficile infection rate | 31 months
  Number of Clostriudium difficile infection cases among all hospital stays included during the study period.
Duration of hospital stay | 31 months
  Number of days during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No